CLINICAL TRIAL: NCT03688295
Title: The Value of Post-operative Antibiotic Therapy After Laparoscopic Appendectomy for Complicated Acute Appendicitis (Other Than for Generalized Peritonitis): a Prospective, Randomized, Placebo-controlled Phase III Study
Brief Title: The Value of Post-operative Antibiotic Therapy After Laparoscopic Appendectomy for Complicated Acute Appendicitis (Other Than for Generalized Peritonitis)
Acronym: ABAP
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI2017_843_0002; 2017-000334-59 (EudraCT Number)
Record Dates: First submitted 2018-06-07; First posted 2018-09-28 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Complicated Acute Appendicitis
Keywords: complicated acute appendicitis; post-operative antibiotic therapy
MeSH Terms: interventions — Anti-Bacterial Agents

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Other): no antibiotherapy post surgery for complicated acute appendicitis (CAA)
  Interventions: Other: No antibiotics
- control group (Active Comparator): antibiotherapy post surgery for complicated acute appendicitis (CAA)
  Interventions: Drug: Antibiotics

INTERVENTIONS:
Other: No antibiotics — Patients will not receive antiobitherapy post surgery for CAA
  Arms: experimental group
Drug: Antibiotics — Patients will receive antiobitherapy post surgery for CAA
  Arms: control group

SUMMARY:
Around 30% of appendectomies are performed for complicated acute appendicitis (CAA, i.e. cases with perforated appendicitis, extraluminal fecaliths, abscesses, or local or generalized peritonitis). The treatment of these complicated forms involves the following steps: initiation of antibiotic treatment at the time of the diagnosis, appendectomy and post-operative antibiotic therapy that continues for 3 days for localized forms of CAA and for 5 days for generalized peritonitis (according to the guidelines issued by the French Society for Anaesthesia and Critical Care Medicine (SFAR)). The results of a Cochrane meta-analysis published in 2005 suggested that the post-operative infection rate was lower in patients having receiving antibiotic therapy after surgery for AA. When only cases of CAA were considered, the difference was no longer significant. However, it should be noted that the studies included in the meta-analysis are now rather old (published before 1995, with open procedures) and no longer provide valid data for answering this question because most appendectomies (80%) are now performed using laparoscopy. Furthermore, a recent cohort study compared a short (3-day) course of antibiotics with a long course (at least 5 days) in patients with CAA having undergone laparoscopic or open appendectomy. There was no significant intergroup difference in the post-operative complication rate. One can thus legitimately question whether post-operative antibiotic therapy is required after laparoscopic appendectomy for CAA.

The purpose of the present study is to evaluate the impact of the absence of post-operative antibiotic therapy on the organ space surgical site infection (SSI) rate in patients presenting with CAA (other than cases of generalized peritonitis) by comparing a group of patients having undergone a conventional strategy of post-operative antibiotic therapy for three days after appendectomy for CAA (the control group) with a group of patients having received a post-operative placebo for three days after appendectomy for CAA (the experimental group). The primary endpoint will be evaluated at one month after randomization.

ELIGIBILITY:
Inclusion Criteria:

1. CAA suspected pre-operatively through a Saint-Antoine score ≤3 and confirmed peroperatively by the presence of a perforated appendicitis, extraluminal fecaliths, abscesses and/or localized peritonitis (pus in one or two abdominal quadrants).
2. Laparoscopic appendectomy.
3. Aged 18 or over
4. Written, informed consent

Exclusion Criteria:

1. Pre-operative exclusion criteria:

   * Patients with cardiac valvulopathy
   * Immunodepressed patients
   * Diabetic patients
   * Patients who have received an antibiotic treatment within 3 months before the surgery (and having a potential impact on the intestinal flora)
   * Related to the diagnosis: other diseases (Crohn's disease, ulcerative colitis, treatment with an immunosuppressive therapy).
   * Related to the severity of the appendicitis:
   * A Saint-Antoine score of 4 or 5 (non-complicated acute appendicitis)
   * Severe sepsis, septic shock, generalized peritonitis
   * Related to the treatment:

     * A decision to perform open appendectomy.
     * Patients who received an adaptive dose of Levofloxacine 250 mg/24H instead of 500 mg/24H in pre-operative or in per-operative (notably for patients with creatinine clearance ≤ 50 ml/min)
     * allergy to metronidazole or to one of the excipient
     * Contra-indication to the use of ceftriaxone (hypersensibility to the active substance, to another cephalosporin, to the excipient of the used speciality), history of severe hypersesibility (as anaphylactic shock), history of hypersensibility to another antibiotic of the beta-lactamin family (penicillin, monobactam, carbapénèmes)
     * Contra-indication to the use of levofloxacin, hypersensibility to levofloxacin, to another quinolone or to the excipient of one of the use speciality, hypersensibility to levofloxacine ou any other quinolone or to any excipient, epilepsia, history of tendinitis when injection of fluoroquinolones.
   * Related to the patient

     * Living at more than one hour from an hospital
     * Patient who has no relative or other third person who could be present at home and provide assistance in case of any problem for the discharged patient
2. Per-operative exclusion criteria (related to the severity of appendicitis):

   * Non-complicated forms (catarrhal appendicitis or the absence of extraluminal fecaliths, abscess or peritonitis).
   * Generalized purulent or stercoral peritonitis (the presence of pus or faeces in more than two quadrants of the abdomen).

In order to assess the reproducibility of the inclusion criteria in the various centres and to avoid variations due to the lack of an official definition for localized peritonitis, all centres will receive a video tutorial on localized peritonitis before the start of the study.

* Pregnancy or breastfeeding.
* Patients under guardianship.
* Patients unable to provide informed consent.
* Patient lacking social security coverage
* Allergy to metronidazole

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1476 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
proportion of patients having developed organ space surgical site infections (SSIs) by postoperative day (POD)30 | postoperative day 30
  primary outcome is the proportion of patients with deep SSIs by POD30. Deep SSIs are officially defined by the CDCcentre of disease control and prevention (CDC) as infections that occur within 30 days of surgery AND appear to be related to the surgery AND affect the organ or the cavity around the surgical site (i.e. any anatomical structure - other than the incision - that is opened or handled during surgery) AND for which at least one of the following signs is observed: pus coming from a drain placed in the organ or cavity; germs isolated from a liquid or tissue sample collected aseptically from the organ or cavity; an abscess or another obvious sign of infection of the organ or cavity found by macroscopic examination during subsequent surgery or in a radiological or histopathological examination.

SECONDARY OUTCOMES:
Quality of life post surgery using the 36-Item Short Form Health Survey | day 0 and day 30
  Quality of life on day 0 and day 30 post surgery, with the 36-Item Short Form Health Survey questionnaires (0 = very bad, 100 = very good)
proportion of patients with superficial SSIs | postoperative day 30
  The proportion of patients with superficial SSIs, defined as infections that occur within 30 days of the intervention AND affect the skin and subcutaneous tissue AND or which at least one of the following signs is observed: pus coming from the superficial part of the incision, germs isolated from a liquid or tissue sample collected aseptically from the superficial part of the incision, a sign of infection (pain, tenderness, redness, burning, etc.) associated with deliberate opening of the superficial part of the incision by the surgeon (except if the culture is negative). Infection of the superficial part of the incision is diagnosed by the surgeon (or the physician attending to the patient).
post-operative infection rates | postoperative day 30
  post-operative infection rates by POD30, including SSIs and remote infections.
number of antibiotic-free days | postoperative day 30
  number of antibiotic-free days between randomization and POD30
Description of the microbial flora | Day 0
  Description of the microbial flora found in the antibiogram of the per-operative sample collected in all cases
balance between antibiotic therapy and microbial resistance | postoperative day 30
  balance between antibiotic therapy and microbial resistance
Evaluation of morbidity and mortality | postoperative day 30
  Evaluation of morbidity and mortality (according to the Dindo-Clavien classification and the Comprehensive Complication Index (CCI)).
Length of hospital stay | postoperative day 30
  Length of hospital stay, defined as the number of days of hospitalization between surgery and discharge
rehospitalization rate | postoperative day 30
  rehospitalization rate, defined as the proportion of patients rehospitalized during the study

CONTACTS AND LOCATIONS:
Locations (1):
- Amiens North Hospital, Amiens, France

REFERENCES:
- [Derived] Sabbagh C, Siembida N, Dupont H, Diouf M, Schmit JL, Boddaert S, Regimbeau JM. The value of post-operative antibiotic therapy after laparoscopic appendectomy for complicated acute appendicitis: a prospective, randomized, double-blinded, placebo-controlled phase III study (ABAP study). Trials. 2020 Jun 1;21(1):451. doi: 10.1186/s13063-020-04411-1. PMID 32487213